CLINICAL TRIAL: NCT00238056
Title: Effect of Domperidone on QT Interval in Premature Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD 05/9-C
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2005-10

CONDITIONS: Prematurity and Feeding Intolerance
Keywords: Domperidone, QT, prematurity
MeSH Terms: conditions — Premature Birth

INTERVENTIONS:
Drug: domperidone Drug

SUMMARY:
30 premature infants treated by domperidone upon decision of the attending neonatologist will have a daily recording of electrocardiogram for the first 7 seven days of treatment, and pharmacokinetics dosages at Day 7. Their ECG will be compared to 30 non treated premature infants, matched for gestational age, postnatal age and sex.

ELIGIBILITY:
Inclusion Criteria:

Gestational age less than 36 weeksPostnatal age greater than 10 days Treated / not treated by domperidone (case/control)Signed parental informed consent

Exclusion Criteria:

Severe cardiac arrhythmia Congenital heart disease (persistent ductus arteriosus excluded)Familial history of congenital long QT syndrome

Min Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Gournay, MD, Principal Investigator — Service de Cardiologie et Service de Réanimation Néonatale CHU de Nantes
Locations (1):
- Centre Hospitalier de Nantes, Nantes, France